CLINICAL TRIAL: NCT04338841
Title: HOME-CoV: Hospitalization or Outpatient ManagEment of Patients With Confirmed or Probable SARS-CoV-2 Infection. A Before and After Implementation of a Consensus Help-decision Making Rule Study
Brief Title: HOME-CoV: Hospitalization or Outpatient ManagEment of Patients With a SARS-CoV-2 Infection
Acronym: HOME-CoV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00831-38
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Infection
Keywords: covid-19; outpatient; expert consensus; decision-making
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Quasi-experimental before and after multicentre prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase1: Before HOME-CoV rule implementation (No Intervention): Observational assessment of current practices: no recommendation is performed.
  Patients consulting Emergency Departments with suspected or probable COVID-19 are evaluated for potential inclusion.
  Clinical, biological and imaging data that may be involved in decision-making about hospitalization are collected as well as the physician final decision (hospitalization or outpatient management) and its main determinants.
  A phone-call follow-up is performed and the clinical status according to the Ordinal Scale for Clinical Improvement of COVID-19 from the World Heath Organization is collected on day 7 and day 28 following inclusion.
- Phase 2: After HOME-CoV rule implementation (Experimental): Observational assessment of practices after implementation of the rule: physicians are recommended to apply the HOME-CoV rule but still free to use other determinants in their decision.
  Patients consulting Emergency Departments with suspected or probable COVID-19 are evaluated for potential inclusion. Clinical, biological and imaging data that may be involved in decision-making about hospitalization are collected as well as the physician final decision (hospitalization or outpatient management) and its main determinants.
  A phone-call follow-up is performed and the clinical status according to the Ordinal Scale for Clinical Improvement of COVID-19 from the World Heath Organization is collected on day 7 and day 28 following inclusion.
  Interventions: Other: HOME-CoV rule implementation

INTERVENTIONS:
Other: HOME-CoV rule implementation — HOME-CoV rule is an easy-to-use clinical rule aiming to help emergency physicians in hospitalisation or outpatient management decision making. The definition of the rule is performed using the Delphi method to reach a consensus of a large panel of experts.
  Between before and after period, educational lectures, posters, and pocket cards showing and explaining HOME-CoV rule are communicated to participating Emergency Departments.
  Arms: Phase 2: After HOME-CoV rule implementation

SUMMARY:
COVID-19 pandemic has developed worldwide in less than 4 months. The clinical presentations are variable widely, ranging from simple rhinitis to major lung damage that can lead to death.

In many countries involved in the ongoing health disaster due to SARS-CoV-2 infection, hospital are overloaded. In this context, the decision to hospitalize or to manage COVID-19 patients at home is crucial and defining reliable and consensual criteria is a major issue.

HOME-CoV study is a multicentre quasi-experimental interventional study, before and after implementation of a help-decision making rule (HOME-CoV rule), developed via the Delphi method.

Our main hypothesis is that a strategy based on the consensual HOME-CoV rule compared to current practice is at least as safe as regards the 7-day-rate of adverse events (safety criterion) and more effective as regards the rate of patients eventually managed as outpatients (efficacy criterion).

DETAILED DESCRIPTION:
Definition of HOME-CoV rule:

The Delphi method is used to reach a consensus of a large panel of experts and to define an easy-to-use clinical rule aiming to help emergency physicians in hospitalisation or outpatient management decision making : the HOME-CoV rule.

The impact of the rule implementation is evaluated in a before and after study:

* before period: observational assessment of current practices
* implementation period : educational lectures, posters, and pocket cards showing and explaining HOME-CoV rule are communicated to participating Emergency Departments.
* after period : observational assessment of practices

In each period, patients consulting Emergency Departments with suspected or probable COVID-19 are evaluated for potential inclusion. Clinical, biological and imaging data that may be involved in decision-making about hospitalization are collected as well as the physician final decision (hospitalization or outpatient management) and its main determinants.

A phone-call follow-up is performed and the clinical status according to the Ordinal Scale for Clinical Improvement of COVID-19 from the World Heath Organization is collected on day 7 and day 28 following inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Admitted for COVID-19 infection confirmed by a positive SARS-CoV2 RT-PCR or considered probable by the physician in charge of the patient.
* Not requiring care in intensive care unit or resuscitation unit or
* No subject of a limitation decision of active therapies,
* Free informed express consent to participate in the study orally given or signed by the patient according to local legislation,
* Insurance cover according to local legislation;

Exclusion Criteria:

* Patient whose main diagnostic hypothesis in the emergency room is not a SARS-CoV-2 infection but another differential diagnosis,
* Patient admitted to the emergency room for 18 hours or more,
* Patient whose follow-up on D28 is impossible, whatever the reason,
* Patient with a poor understanding of the French language,
* Patient already included in the study,
* Person deprived of their liberty by judicial or administrative decision,
* Person under psychiatric care under duress,
* Person subject to a legal protection measure,
* Person unable to express consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3133 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
the composite rate of adverse outcomes | day 7
  Adverse outcomes include intubation with mechanical ventilation requirement and death (Stage ≥ 6 on "Ordinal Scale for Clinical Improvement" of the World Health Organization) within 7 days after inclusion.
The rate of hospitalization | 24 hours
  The rate of patients hospitalized after admission to the emergency room including patients discharged home more than 24 hours after admission.
  It will be analyzed in a hierarchical approach, only if first primary objective is positive i.e. non-inferiority of HOME-CoV strategy versus current practice on the rate of adverse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine DOUILLET, Principal Investigator — University Hospital, Angers
Locations (29):
- Belgium (2):
  - Clinique Universitaire Saint-Luc, Brussels
  - CHU de Liège, Liège
- France (26):
  - Ch Argenteuil, Argenteuil
  - CH Cholet, Cholet
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Ch Colmar, Colmar
  - CH Alpes Lemant, Contamine-sur-Arve
  - CHU Dijon, Dijon
  - CH Le Mans, Le Mans
  - CH Libourne, Libourne
  - CH Limoges, Limoges
  - Ch Longjumeau, Longjumeau
  - Chu Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - CH Niort, Niort
  - Hopital Paris Saint Joseph, Paris
  - Hopital Saint Antoine, Paris
  - Hôpital Bichat, Paris
  - Hôpital Lariboisière, Paris
  - CHU de Poitiers, Poitiers
  - CH Reims, Reims
  - Ch Remiremont, Remiremont
  - Chu Rennes, Rennes
  - CHU de Rouen, Rouen
  - CH de Saint-Brieuc, Saint-Brieuc
  - CHU de St Etienne, Saint-Etienne
  - Ch Troyes, Troyes
  - CH VICHY, Vichy
- CH Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Douillet D, Penaloza A, Mahieu R, Morin F, Chauvin A, Gennai S, Schotte T, Montassier E, Thiebaud PC, Ghuysen Francois A, Dall'acqua D, Benhammouda K, Bissokele P, Violeau M, Joly LM, Andrianjafy H, Soulie C, Savary D, Riou J, Roy PM; Hospitalization or Outpatient Management of Patients With SARS-CoV-2 Infection Study Group. Outpatient Management of Patients With COVID-19: Multicenter Prospective Validation of the Hospitalization or Outpatient Management of Patients With SARS-CoV-2 Infection Rule to Discharge Patients Safely. Chest. 2021 Oct;160(4):1222-1231. doi: 10.1016/j.chest.2021.05.008. Epub 2021 May 15. PMID 34004154
- [Derived] Douillet D, Mahieu R, Boiveau V, Vandamme YM, Armand A, Morin F, Savary D, Dubee V, Annweiler C, Roy PM; HOME-CoV expert group. Outpatient management or hospitalization of patients with proven or suspected SARS-CoV-2 infection: the HOME-CoV rule. Intern Emerg Med. 2020 Nov;15(8):1525-1531. doi: 10.1007/s11739-020-02483-0. Epub 2020 Sep 4. PMID 32888112